CLINICAL TRIAL: NCT00960830
Title: Mirtazapine Reduces ICD Appropriate Shocks in Cardioverter Implanted Patients With Depression and Anxiety
Brief Title: Mirtazapine Reduces ICD Shocks in ICD Patients With Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Rosario (Other)
Responsible Party: daniel serrani, facultad de psicologia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: PS990
Record Dates: First submitted 2009-07-21; First posted 2009-08-18 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mirtazapine (Placebo Comparator)
  Interventions: Drug: mirtazapine
- mirtazapine, sugar pill (Placebo Comparator)
  Interventions: Drug: mirtazapine

INTERVENTIONS:
Drug: mirtazapine — mirtazapine 15 mg daily tablets
  Other Names: mirtazapine 1500 mtz
  Arms: mirtazapine
Drug: mirtazapine — 15 mg daily
  Other Names: remeron 1569 rem

SUMMARY:
The purpose of this study is to evaluate if the use of antidepressant medication in depressed patients with implantable cardioverter defibrillator reduces the number of ICD's shocks as it improves depressive affect.

DETAILED DESCRIPTION:
episodes of arrhythmia remain present even after icd implantation, this is specially true in depressed patients. it is hypothesized that improving mood state by means of an antidepressant drug . namely mirtazapine. could be responsible of alleviating the number of appropriate shocks delivered by the cardioverter. this could be due to a direct effect of the drug itself or an indirect effect of improving anxious and depressive affect. the mood and anxiety state are measured with the HADS scale

ELIGIBILITY:
Inclusion Criteria:

* cardioverter implanted patients
* depression
* anxiety

Exclusion Criteria:

* heart failure
* other diseases reducing physical fitness

Ages: 65 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
number of implantable cardioverter defibrillator shocks | one year

SECONDARY OUTCOMES:
improvement of depression | one year

CONTACTS AND LOCATIONS:
Overall Officials: daniel jl serrani, MD, Principal Investigator — facultad de psicologia
Locations (1):
- Cl Sn Nicol, San Nicolás, Bs As, Argentina